CLINICAL TRIAL: NCT01272713
Title: A Randomised Controlled Trial of Oxygen Therapy in Acute Myocardial Infarction (AVOID - Air Verses Oxygen In myocarDial Infarction Study)
Brief Title: Air Verses Oxygen In myocarDial Infarction Study
Acronym: AVOID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Ambulance Victoria (Other Government); Monash University (Other); Baker Heart and Diabetes Institute (Other); FALCK Foundation (Unknown)
Responsible Party: Principal Investigator, Ms. Rowan Frew, A.Professor Stephen Bernard, Bayside Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC/10/ALFRED/52
Record Dates: First submitted 2010-12-22; First posted 2011-01-10 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxygen therapy (Other): * Standard acute coronary syndrome treatment as per hospital protocol
  * Pre-hospital supplemental oxygen administered via Hudson mask at a flow rate of 8L/min
  * In-hospital oxygen as per hospital protocol
  Interventions: Other: Oxygen therapy
- No oxygen therapy (Other): * Standard acute coronary syndrome treatment as per hospital protocol
  * No oxygen pre-hospital or in-hospital unless the oxygen saturation falls below 94% in which case oxygen will be administered via nasal cannulae (4L/min) or Hudson mask (8L/min) and titrated to achieve oxygen saturation of 94%.
  Interventions: Other: No oxygen therapy

INTERVENTIONS:
Other: Oxygen therapy — * Pre-hospital supplemental oxygen administered via Hudson mask at a flow rate of 8L/min
  * In-hospital oxygen as per hospital protocol
  Arms: Oxygen therapy
Other: No oxygen therapy — No oxygen pre-hospital or in-hospital unless the oxygen saturation falls below 94% in which case oxygen will be administered via nasal cannulae (4L/min) or Hudson mask (8L/min) and titrated to achieve oxygen saturation of 94%.
  Arms: No oxygen therapy

SUMMARY:
- Aim

The AVOID (Air Verses Oxygen In myocardial infarction) trial is designed to determine if the withholding of routine oxygen therapy in patients with acute heart attack leads to reduced heart damage compared to the current practice of routine inhaled oxygen for all patients.

- Background

There is evidence supporting and refuting the current practice of providing oxygen to all patients with acute heart attack. A recent summary of clinical trials suggested that oxygen may increase the degree of heart damage during heart attack. It also highlighted that the few trials into oxygen therapy were performed before the use of modern medications and procedures to treat heart attack and that further studies were urgently needed, using contemporary practices.

- Design

A total of 334 patients will participate in this randomized controlled trial. Patients in this study will receive the best current management and care for their condition. Patients will be randomized to routine pre-hospital care with oxygen therapy vs pre-hospital care without oxygen therapy. Patients will then receive standard hospital care, aside from allocated oxygen or no oxygen therapy. The primary outcome measure of heart damage will be investigated using routine blood tests. With additional information gathered from other aspects of routine heart care including coronary angiogram, electrocardiograms and complications of hospital stay. Patients will be followed up at 6 months to determine any longer term effects of treatment.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a leading cause of morbidity and mortality in Australia[1]. In particular, many patients with CAD present with ST-elevation myocardial infarction (STEMI) as a result of acute thrombotic coronary artery occlusion. The optimal treatment for patients presenting with STEMI is reperfusion therapy either with primary percutaneous coronary intervention (PCI) or administration of a thrombolytic drug[2, 3].

Current guidelines recommend additional treatments for patients with STEMI prior to reperfusion therapy, such as oxygen, aspirin and nitrates[4]. Whilst there is supportive evidence from clinical trials for the administration of aspirin[5] and nitrates[6], there is no data from prospective, randomised, controlled clinical trials to support the use of routine supplemental oxygen.

For many years, the administration of supplemental oxygen has been considered beneficial for the treatment of patients with acute myocardial infarction largely based on experimental laboratory data. For example, in a laboratory study, anaesthetised dogs underwent coronary artery occlusion and were then administered either 21% oxygen, 40% oxygen or 100% oxygen. In the 40% oxygen group, there was decreased myocardial injury and infarct size compared with the air or 100% oxygen groups[7].

In another laboratory study, two groups of dogs underwent 90 minutes of coronary occlusion followed by 72 hours of reperfusion[8]. One group received 100% inspired oxygen from 20 minutes before reperfusion and three hours after reperfusion whereas the air group received room air. The infarct size in the oxygen group was reduced by 38% and left ventricular ejection fraction was improved compared with the dogs receiving room air. This data suggests that high concentrations of inspired oxygen may be of benefit in acute myocardial infarction followed by reperfusion therapy.

However, there is increasing clinical data that suggests that oxygen administration before and during reperfusion in patients with STEMI may be harmful.

For example, the hemodynamic effects of inhalation of oxygen in high concentration has been investigated in 50 patients with acute myocardial infarction[9]. This resulted in adverse effects including a fall in cardiac output, a rise in blood pressure and an increase systemic vascular resistance. The latter would be expected to increase myocardial work and increase myocardial ischaemia.

There have been three prospective, controlled trials of supplemental oxygen compared with no supplemental oxygen in patients with myocardial infarction.

In a double-blind, randomised in-hospital study, two-hundred patients with myocardial infarction were allocated to receive supplemental oxygen or air administered by face mask for the initial 24 hours in hospital[10]. The two groups were comparable at baseline. There was no significant difference in mortality, incidence of arrhythmias or use of analgesics between the groups. There was a higher incidence of sinus tachycardia in the patients given oxygen. This study suggested that there was no benefit from the routine administration of oxygen in uncomplicated myocardial infarction.

In a second study, 50 patients were allocated to either supplemental oxygen or room air[11]. The main outcome measure was the requirement for analgesia with 16 of 22 patients (72.7%) in the oxygen group using opiates for pain relief compared with 18 of 20 patients (90%) in the air group. This study did not report mortality rate.

In a third study conducted in Russia, 137 patients were allocated to either supplemental oxygen (4-6L/Min) or air[12]. Complications including heart failure, pericarditis and rhythm disorders occurred less frequently in the air group (Risk ratio 0.45: 95% CI 0.22 to 0.94). One patient out of 58 died in the oxygen group and none out of 79 participants in the air group.

A meta-analysis analysed the outcomes in the 387 patients included in these three studies[13]. The pooled risk ratio of death for patients allocated to oxygen administration was 2.88 (95% CI 0.88 to 9.39) in an intention-to-treat analysis and 3.03 (95% CI 0.93 to 9.83) in patients with confirmed myocardial infarction. While suggestive of harm, the small number of deaths recorded meant that this finding did not reach statistical significance. Pain was measured by analgesic use and the pooled risk ratio for decreased use of analgesics in the oxygen group was 0.97 (95% CI 0.78 to 1.20).

In addition to the above studies, other clinical studies have examined the use of novel techniques for additional oxygen delivery to the ischemic myocardium during reperfusion. In a clinical trial testing the role of hyperbaric oxygen (HBO) in myocardial infarction, 112 patients with STEMI were allocated to either HBO or usual supplemental oxygen (40% by mask or 6L/min by nasal prongs) during thrombolysis[14]. There was no significant difference between the groups in creatinine kinase levels at 24 hours or left ventricle ejection fraction (LVEF) on discharge. Overall, there was no overall benefit with this approach found in this study.

In a clinical trial testing coronary artery reperfusion with hyperoxic blood during reperfusion, 269 patients with acute AMI undergoing PCI were randomly assigned to receive hyperoxemic blood reperfusion or normoxemic blood reperfusion by catheter into the area of reperfused myocardium[15]. At 30 days, there was no significant difference in the infarct size, ST-segment resolution, or regional wall motion score. Although improvement in cardiac function was seen in patients with anterior MI who were reperfused within 6 hours, this finding was a post-hoc analysis.

A meta-analysis of all studies of hyperoxic myocardial reperfusion found that this treatment caused a significant reduction in coronary blood flow, an increase in coronary vascular resistance and a significant reduction in myocardial oxygen consumption[16]. This data appears to confirm that supplemental oxygen may be harmful.

Given the lack of clinical data of the efficacy of oxygen administration, European guidelines for the management of acute coronary syndromes do not now include a recommendation for supplemental oxygen[17]. Whilst the recent American Heart Association guideline for the management of acute coronary syndromes does recommend oxygen, they note that there is no clinical trial evidence to support this recommendation[4]. The most recent addendum to the 2006 Australian National Heart Foundation Guidelines does not recommend the routine use of supplemental oxygen[18].

In summary, whilst there is some laboratory evidence of benefit for supplemental oxygen during STEMI and reperfusion, the available clinical data suggests that oxygen may be of no use or even harmful. Since oxygen is currently used routinely in many ambulance services and hospitals in the treatment of acute coronary syndromes, prospective clinical trials comparing supplemental oxygen with no supplemental oxygen in this condition are required[19, 20].

Ambulance Victoria is uniquely placed to undertake this research. The Mobile Intensive Care Ambulances (MICA) of Ambulance Victoria are equipped with 12 lead ECG capability and pulse-oximetry monitors. In Melbourne, MICA attends approximately 400 STEMI patients per year.

We therefore propose to undertake a randomised, controlled trial comparing supplemental oxygen therapy with air in patients without hypoxia who present with STEMI to determine the effect on the size of the myocardial infarct at hospital discharge.

- References

1. AIHW. Australian Institute of Health and WelfareCardiovascular disease mortality: trends at different ages. Cardiovascular series no 31 Cat no47 Canberra: AIHW 2010.
2. Antman EM, Anbe DT, Armstrong PW, et al. ACC/AHA Guidelines for the Management of Patients With ST-Elevation Myocardial Infarction. Circulation 2004;110:e82-293.
3. Guidelines for the management of acute coronary syndromes 2006. Med J Aust 2006;184:S9-29.
4. O'Connor RE, Brady W, Brooks SC, et al. Part 10: Acute Coronary Syndromes: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation 2010;122:S787-817.
5. Freimark D, Matetzky S, Leor J, et al. Timing of aspirin administration as a determinant of survival of patients with acute myocardial infarction treated with thrombolysis. Am J Cardiol 2002;89:381-5.
6. Charvat J, Kuruvilla T, al Amad H. Beneficial effect of intravenous nitroglycerin in patients with non-Q myocardial infarction. Cardiologia 1990;35:49-54.
7. Maroko PR, Radvany P, Braunwald E, Hale SL. Reduction of infarct size by oxygen inhalation following acute coronary occlusion. Circulation 1975;52:360-8.
8. Kelly RF, Hursey TL, Parrillo JE, Schaer GL. Effect of 100% oxygen administration on infarct size and left ventricular function in a canine model of myocardial infarction and reperfusion. Am Heart J 1995;130:957-65.
9. Kenmure ACF, Murdoch WR, Beattie AD, Marshall JCB, Cameron AJV. Circulatory and Metabolic Effects of Oxygen in Myocardial Infarction. Br Med J 1968;4:360-4.
10. Rawles JM, Kenmure AC. Controlled trial of oxygen in uncomplicated myocardial infarction. Br Med J 1976;1:1121-3.
11. Wilson AT, Channer KS. Hypoxaemia and supplemental oxygen therapy in the first 24 hours after myocardial infarction: the role of pulse oximetry. J R Coll Physicians Lond 1997;31:657-61.
12. Ukholkina GB, Kostianov I, Kuchkina NV, Grendo EP, Gofman Ia B. [Effect of oxygenotherapy used in combination with reperfusion in patients with acute myocardial infarction]. Kardiologiia 2005;45:59.
13. Cabello JB, Burls A, Emparanza JI, Bayliss S, Quinn T. Oxygen therapy for acute myocardial infarction. Cochrane Database Syst Rev 2010;6:CD007160.
14. Stavitsky Y, Shandling AH, Ellestad MH, et al. Hyperbaric oxygen and thrombolysis in myocardial infarction: the 'HOT MI' randomized multicenter study. Cardiology 1998;90:131-6.
15. O'Neill WW, Martin JL, Dixon SR, et al. Acute Myocardial Infarction With Hyperoxemic Therapy (AMIHOT): A Prospective, Randomized Trial of Intracoronary Hyperoxemic Reperfusion After Percutaneous Coronary Intervention. Journal of the American College of Cardiology 2007;50:397-405.
16. Farquhar H, Weatherall M, Wijesinghe M, et al. Systematic review of studies of the effect of hyperoxia on coronary blood flow. American Heart Journal 2009;158:371-7.
17. Bassand J-P, Hamm CW, Ardissino D, et al. Guidelines for the diagnosis and treatment of non-ST-segment elevation acute coronary syndromes. European Heart Journal 2007;28:1598-660.
18. ACS writing group. 2010 addendum to the National Heart Foundation of Australia/Cardiac Society of Australia and New Zealand guidelines for the management of acute coronary syndromes (ACS) 2006. Final Draft form 2010.
19. Wijesinghe M, Perrin K, Ranchord A, Simmonds M, Weatherall M, Beasley R. Routine use of oxygen in the treatment of myocardial infarction: systematic review. Heart 2009;95:198-202.
20. Moradkhan R, Sinoway LI. Revisiting the Role of Oxygen Therapy in Cardiac Patients. J Am Coll Cardiol 2010;56:1013-6.
21. Di Chiara A, Dall'Armellina E, Badano LP, Meduri S, Pezzutto N, Fioretti PM. Predictive value of cardiac troponin-I compared to creatine kinase-myocardial band for the assessment of infarct size as measured by cardiac magnetic resonance. Journal of Cardiovascular Medicine 2010;11:587-92 10.2459/JCM.0b013e3283383153.
22. Chia S, Senatore F, Raffel OC, Lee H, Wackers FJT, Jang I-K. Utility of Cardiac Biomarkers in Predicting Infarct Size, Left Ventricular Function, and Clinical Outcome After Primary Percutaneous Coronary Intervention for ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol Intv 2008;1:415-23.
23. Hallén J, Maria S, Per J, Dan A, Peter MC. Influence of ST-Segment Recovery on Infarct Size and Ejection Fraction in Patients With ST-Segment Elevation Myocardial Infarction Receiving Primary Percutaneous Coronary Intervention. The American Journal of Cardiology 2010;105:1223-8.
24. Gotberg M, Olivecrona GK, Koul S, et al. A Pilot Study of Rapid Cooling by Cold Saline and Endovascular Cooling Before Reperfusion in Patients With ST-Elevation Myocardial Infarction. Circ Cardiovasc Interv 2010:CIRCINTERVENTIONS.110.957902.
25. Wright J, Adriaenssens T, Dymarkowski S, Desmet W, Bogaert J. Quantification of Myocardial Area at Risk With T2-Weighted CMR: Comparison With Contrast-Enhanced CMR and Coronary Angiography. JACC: Cardiovascular Imaging 2009;2:825-31.
26. Roubille F, Samri A, Cornillet L, et al. Routinely-feasible multiple biomarkers score to predict prognosis after revascularized STEMI. European journal of internal medicine 2010;21:131-6.
27. Davis DP, Graydon C, Stein R, et al. The Positive Predictive Value of Paramedic Versus Emergency Physician Interpretation of the Prehospital 12-Lead Electrocardiogram. Prehospital Emergency Care 2007;11:399-402.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* Chest pain for < 12 hours
* ST-elevation Myocardial Infarction including either: 1) Persistent ST-segment elevation of ≥1mm in two contiguous limb leads; 2) ST-segment elevation of ≥ 2mm in two contiguous chest leads, or; 3) New left bundle branch block (LBBB) pattern.
* Able to be transported to a participating hospital

Exclusion Criteria:

* Hypoxia with oxygen saturation measured on pulse oximeter < 94% with the patient breathing air
* Bronchospasm requiring nebulised salbutamol therapy using oxygen
* Altered conscious state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Myocardial Infarct Size | At 72 hours post infarct
  The primary end-point for the study will be infarct size at hospital discharge which will be ascertained by the routinely collected cardiac biomarkers during hospital admission such as cardiac troponin I (cTnI) and creatine kinase (CK)Infarct size will be evaluated via blood test on admission and then 6 hourly tests for 48 hours and 12 hourly measurements between 48 hours and 72 hours. Infarct size will be measured by:
  * Mean and peak cTnI
  * Mean and peak CK
  * The area under the curve of CK and cTnI release over the first 72 hours of reperfusion.

SECONDARY OUTCOMES:
ST segment resolution | 1 day post reperfusion
TIMI Flow | At completion of coronary intervention procedure
  TIMI - Thrombolysis in Myocardial infarction score
Survival to Hospital Discharge | Any
Major Adverse Cardiac Events (MACE) | 6 months
  Death, recurrent myocardial infarction, and re-hospitalization measured at 6 months
Myocardial Salvage | 4 days and 6 months
  Magnetic resonance imaging (MRI) measurement of infarct size as percent of area at risk determined with T2-weighted MRI (in small sub set of patients) at day 4 and repeated at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bernard, MBBS MD, Principal Investigator — Alfred Hospital, Monash University, Ambulance Victoria; Karen Smith, BSc PhD, Principal Investigator — Ambulance Victoria, Monash University; Dion Stub, MBBS, Study Director — Alfred Hospital, Baker IDI Institute, Monash University; Ian Meredith, BSc MBBS PhD, Study Director — Southern Health, Monash University; Michael Stephenson, RN BA, Study Director — Ambulance Victoria; Janet Bray, RN PhD, Study Director — Ambulance Victoria; Bill Barger, ADHS, Study Director — Ambulance Victoria; David Kaye, MBBS PhD, Study Director — Alfred Hospital, Baker IDI Institute, Monash University; Peter Cameron, MBBS MD, Study Director — Alfred Hospital, Monash University
Locations (10):
- Australia (10):
  - Peninsula Private Hospital, Frankston, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Western Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincents Hospital, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Ambulance Victoria, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Frankston Hospital, Melbourne, Victoria

REFERENCES:
- [Background] Stub D, Smith K, Bernard S, Bray JE, Stephenson M, Cameron P, Meredith I, Kaye DM; AVOID Study. A randomized controlled trial of oxygen therapy in acute myocardial infarction Air Verses Oxygen In myocarDial infarction study (AVOID Study). Am Heart J. 2012 Mar;163(3):339-345.e1. doi: 10.1016/j.ahj.2011.11.011. PMID 22424003
- [Derived] Stub D, Smith K, Bernard S, Nehme Z, Stephenson M, Bray JE, Cameron P, Barger B, Ellims AH, Taylor AJ, Meredith IT, Kaye DM; AVOID Investigators. Air Versus Oxygen in ST-Segment-Elevation Myocardial Infarction. Circulation. 2015 Jun 16;131(24):2143-50. doi: 10.1161/CIRCULATIONAHA.114.014494. Epub 2015 May 22. PMID 26002889